CLINICAL TRIAL: NCT04750577
Title: Randomised, Double-blind (Within Dose Groups), Placebo-controlled and Parallel Group Trial to Investigate the Effects of Different Doses of Oral BI 685509 Given Over 20 Weeks on UACR Reduction in Patients With Diabetic Kidney Disease
Brief Title: A Study to Test the Effect of Different Doses of BI 685509 on Kidney Function in People With Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1366-0005; 2020-002929-28 (EudraCT Number)
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-blind (within dose groups), parallel, placebo-controlled trial. Patients will be randomised equally into one of three parallel dose groups, and in each dose group to treatment either with BI 685509 or matching placebo in a 3:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 685509
- BI 685509 1 mg TID (Experimental)
  Interventions: Drug: BI 685509
- BI 685509 2 mg TID (Experimental): Low dose followed by up-titration to medium dose.
  Interventions: Drug: BI 685509
- BI 685509 3 mg TID (Experimental): Low dose followed by up-titration to medium dose, followed by up-titration to high-dose.
  Interventions: Drug: BI 685509

INTERVENTIONS:
Drug: Placebo matching BI 685509 — film-coated tablet
  Arms: Placebo
Drug: BI 685509 — film-coated tablet
  Other Names: Avenciguat
  Arms: BI 685509 1 mg TID; BI 685509 2 mg TID; BI 685509 3 mg TID

SUMMARY:
This study is open to adults with diabetic kidney disease. The purpose of the study is to find out whether a medicine called BI 685509 improves kidney function. Three different doses of BI 685509 are tested in this study.

Participants get either one of the three doses of BI 685509 or placebo. It is decided by chance who gets which BI 685509 dose and who gets placebo. Participants take BI 685509 or placebo as tablets 3 times a day. Placebo tablets look like BI 685509 tablets but do not contain any medicine. Participants continue taking their usual medicine for diabetes and kidney disease throughout the study.

Participants are in the study for about 7 months. During this time, they visit the study site about 11 times. Where possible, about 6 of the 11 visits can be done at the participant's home instead of the study site. The trial staff may also contact the participants by phone or video call.

Kidney function is assessed based on the analysis of urine samples, which participants collect at home. At the end of the trial the results are compared between the different doses of BI 685509 and placebo. During the study, the doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent in accordance with International Council of Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
2. Male or female patients aged ≥ 18 years at time of consent.
3. eGFR (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 20 and < 90 mL/min/1.73 m2 at Visit 1 by central laboratory analysis. eGFR must remain ≥ 20 mL/min/1.73 m2 after Visit 1 up to the start of Visit 3, measured by central or any local laboratory analysis.
4. Urine Albumin Creatinine Ratio (UACR) ≥ 200 and < 3,500 mg/g in spot urine (midstream urine sample) by central laboratory analysis at Visit 1.
5. Treatment with the highest tolerated dose of either Angiotensin Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) (but not both together), and stable dose for ≥ 4 weeks before Visit 1 with no planned change of the therapy during the trial.
6. If the patient is taking any of the following medications they should be on a stable dose at least 4 weeks prior to visit 1 until start of treatment, with no planned change of the therapy during the trial: anti-hypertensives, Non-steroidal anti-inflammatory drug(s) (NSAIDs), endothelin receptor antagonists, systemic steroids or Sodium-Glucose co-Transporter-2 (SGLT2) inhibitors.
7. Patients with stable type 1 or type 2 diabetes mellitus, diagnosed before informed consent. Treatment (including SGLT2 inhibitor and/or Glucagon-Like Peptide 1 (GLP1) receptor agonist) should have been unchanged or changes deemed minor (according to investigator's judgement) within 4 weeks before Visit 1 and until start of trial treatment.
8. Glycated Haemoglobin (HbA1c) < 10.0% at Visit 1 measured by the central laboratory.

Further inclusion criteria apply.

Exclusion criteria:

1. Treatment with Renin Angiotensin Aldosterone System (RAAS) interventions (apart from either ACEi or ARB), phosphodiesterase 5 inhibitors, non-specific phosphodiesterase inhibitors (such as dipyridamole and theophylline), NO donors including nitrates, sGC-stimulators/activators (other than trial treatment) or any other restricted medication (including OATP1B1/3 inhibitors, UGT inhibitors/inducers) as provided in the Investigator Site File (ISF) within 4 weeks prior to visit 1 and throughout screening and baseline run-in. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial are also excluded.
2. Any clinically relevant laboratory value from screening until start of trial treatment, which in the investigator's judgement puts the patient at additional risk.
3. Biopsy or otherwise confirmed non-diabetic chronic kidney disease, or non-diabetic chronic kidney disease in the opinion of investigator, e.g., Autosomal Dominant Polycystic Kidney Disease (ADPKD), uncontrolled lupus nephritis. The presence of a hypertensive etiology does not need to be excluded unless it is evident this is the only cause for the Chronic Kidney Disease (CKD).
4. Any immunosuppression therapy or immunotherapy in the last 3 months prior to visit 1 and throughout screening and baseline run-in (except prednisolone ≤10 mg or equivalent).
5. Acute kidney injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) in the 30 days prior to Visit 1 until the start of trial treatment.
6. Planned start of chronic renal replacement therapy during the trial or end stage renal disease before start of trial treatment.
7. Known history of moderate or severe symptomatic orthostatic dysregulation as judged by the investigator before start of trial treatment.
8. The patient has an active infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) (or is known to have a positive test) from screening until randomisation.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (17):
  - Kidney & Hypertension Center, Victorville, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Indago Research and Health Center, Hialeah, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Davita Clinical Research, Columbus, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Research by Design, LLC, Chicago, Illinois
  - DaVita Clinical Research, Las Vegas, Nevada
  - Total Renal Research, The Bronx, New York
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - DaVita Clinical Research, Houston, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - DaVita Clinical Research, San Antonio, Texas
  - Kidney Specialists of North Houston, PLLC, Shenandoah, Texas
  - Tidewater Kidney Specialists, Norfolk, Virginia
- Argentina (6):
  - CEDIC - Centro de Investigacion Clinica, CABA
  - Instituto Médico Especializado, Capital Federal
  - Instituto Privado de Investigaciones Clínica Córdoba S.A., Córdoba
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto Médico Catamarca - IMEC, Rosario
  - CEREHA S.A.- Centro de Estudios Renales e Hipertensión Arterial, Sarandí
- Australia (6):
  - Renal Research, Gosford, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Austin Health, Heidelberg, Victoria
- Canada (3):
  - CARe Clinic, Red Deer, Alberta
  - Albion Finch Medical Centre, Toronto, Ontario
  - Fadia El Boreky Medicine Professional, Waterloo, Ontario
- China (4):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - People's Hospital of Sichuan Province, Sichuan
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Steno Diabetes Center Copenhagen, Herlev
  - Sjællands Universitetshospital, Roskilde
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong
- Japan (12):
  - Chubu Rosai Hospital, Aichi, Nagoya
  - Daido Hospital, Aichi, Nagoya
  - Kurume University Hospital, Fukuoka, Kurume
  - Nakayamadera Imai Clinic, Hyogo, Takarazuka
  - Takai Naika Clinic, Kanagawa, Kamakura
  - Kawasaki Medical School Hospital, Okayama, Kurashiki
  - Osaka General Medical Center, Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - ToCROM Clinic, Tokyo, Shinjyuku-ku
- Malaysia (4):
  - University Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Universiti Sains Malaysia Hospital, Kelantan
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
- Mexico (4):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Clinstile S.A. de C.V., México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Netherlands (2):
  - Albert SchweitzerZiekenhuis, Dordrecht
  - Universitair Medisch Centrum Utrecht, GA Utrecht
- New Zealand (2):
  - P3 Research Kapiti, Paraparaumu
  - P3 Research, Tauranga
- Poland (4):
  - SPECDERM Poznanska General Partnership, Bialystok
  - Pratia MCM Krakow, Krakow
  - Medicome Limited Liability Company, Oświęcim
  - NBR Polska, Warsaw
- Portugal (2):
  - ULS da Região de Aveiro, Aveiro
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
- Spain (4):
  - Hospital A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Virgen Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
- United Kingdom (2):
  - University Hospital Coventry, Coventry
  - Barts and The London School of Medicine and Dentistry, London

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Heerspink HJL, Cherney D, Gafor AHA, Gorriz JL, Pergola PE, Tang SCW, Desch M, Iliev H, Sun Z, Steubl D, Nangaku M. Effect of Avenciguat on Albuminuria in Patients with CKD: Two Randomized Placebo-Controlled Trials. J Am Soc Nephrol. 2024 Sep 1;35(9):1227-1239. doi: 10.1681/ASN.0000000000000418. Epub 2024 May 25. PMID 38795055
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a phase II, randomized, double-blind (within dose groups), placebo controlled and parallel group trial in patients with diabetic kidney disease (DKD) to demonstrate the effectiveness of BI 685509 and to characterize the dose-response relationship for BI 685509 in patients with DKD by assessing 3 doses and placebo.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 685509 1 mg TID: The patients were administered 1 milligram (mg) BI 685509 Film-coated tablets 3 times a day during 20 weeks of treatment in total, with water and taken with or without food. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- BI 685509 2mg TID: The patients were administered 1 milligram (mg) BI 685509 Film-coated tablets 3 times a day during the first 2 weeks of treatment, If the medication was tolerated, up-titration to 2 mg TID BI 685509 occurred after 2 weeks until Week 20 of treatment. The tablets were taken with water, with or without food. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- BI 685509 3 mg TID: The patients were administered 1 milligram (mg) BI 685509 Film-coated tablets 3 times a day during the first 2 weeks of treatment, If the medication was tolerated, up-titration to 2 mg TID BI 685509 occurred after 2 weeks until Week 4 of treatment. Then if medication was tolerated, up-titration to 3 mg TID BI 685509 occurred from Week 5 until Week 20.
  The tablets were taken with water, with or without food. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- Placebo: This arm comprises all placebo treated participants. Participants were randomized in the dose group in a 3:1 ratio (test treatment to placebo). Participants were administered Film-coated tablets of matching placebo 3 times a day during 20 weeks of treatment. The tablets were taken with water, with or without food. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo
Started (Randomised) | 61 | 61 | 61 | 60
Treated | 61 | 61 | 61 | 58
Completed | 55 | 46 | 47 | 53
Not Completed | 6 | 15 | 14 | 7
Not completed — Adverse Event | 2 | 10 | 8 | 1
Not completed — Change of residence | 0 | 0 | 1 | 0
Not completed — Burden of study procedures | 0 | 2 | 2 | 0
Not completed — Prematurely discontinued | 0 | 0 | 0 | 2
Not completed — Protocol deviation | 1 | 1 | 1 | 1
Not completed — Other than listed | 3 | 2 | 2 | 1
Not completed — Not treated | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): This patient set includes all entered and randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo | Total
Number analyzed (Participants) | 61 | 61 | 61 | 60 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (9.3) | 64.8 (11.0) | 65.2 (8.8) | 67.6 (8.7) | 65.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 13 | 16 | 59
  Male | 45 | 47 | 48 | 44 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 23 | 21 | 81
  Not Hispanic or Latino | 45 | 40 | 38 | 39 | 162
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 3 | 2 | 9
  Asian | 23 | 16 | 16 | 16 | 71
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 6 | 11 | 10 | 6 | 33
  White | 30 | 31 | 32 | 34 | 127
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Urine Albumin Creatinine Ratio (UACR) FMV [Mean (Standard Deviation); unit: Milligram/gram (mg/g)] — Urine Albumin Creatinine Ratio (UACR) at baseline. The first morning void (FMV) is the first urination after the patient wakes up at their usual time to start their day. Baseline is defined as the mean of all available samples prior to Visit 2 up to and including those prior to the first intake of trial medication.
  Milligram/gram (mg/g) | 991.7 (889.0) | 1033 (760.4) | 818.4 (686.9) | 866.1 (658.1) | 927.5 (754.8)
Urine Albumin Creatinine Ratio (UACR) - 10 Hour [Mean (Standard Deviation); unit: milligram/gram (mg/g)] — Urine Albumin Creatinine Ratio (UACR) at baseline. For 10-hour urine. Baseline was defined as the mean of all non-missing assessments from visit 2 until prior to the first intake of trial medication. As soon as the First Morning Void sample was collected the clock starts for the 10-hour urine collection. During the 10-hour period every time the patient urinates, they collected their urine into a provided container. An aliquot of this urine was taken and used as the 10-hour UACR sample.
  milligram/gram (mg/g) | 1093.5 (980.3) | 1090.7 (794.4) | 880.8 (722.4) | 913.1 (657.3) | 994.9 (799.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log Transformed Urine Albumin Creatinine Ratio (UACR) Measured in 10-hour Urine After 20 Weeks of Trial Treatment
Description: Change from baseline in log transformed Urine Albumin Creatinine Ratio (UACR) after 20 weeks is reported. As soon as the First Morning Void sample was collected the clock starts for the 10-hour urine collection. During the 10-hour period every time the patient urinates, they collected their urine into a provided container. An aliquot of this urine was taken and used as the 10-hour UACR sample. Least Square Means and Standard error were estimated by restricted maximum likelihood based Mixed-effect Model for Repeated Measures ((REML)-based MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12 and Week 20) as well as random effects of patient. The Least Squares Mean (Standard error) at Week 20 is reported.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated UACR measurements from baseline (Week -2 and Week -1) and Week 6, Week 12 and Week 20. The data represent the Least Squares Mean at Week 20.
Population: Full Analysis Set (FAS): The patient set included all patients who had at least one baseline measurement of UACR in week -2, -1, or 0 and at least one post-baseline measurement after week 6.
Measure: Least Squares Mean (Standard Error); unit: milligram/gram (mg/g)
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo
Number analyzed (Participants) | 57 | 53 | 56 | 56
milligram/gram (mg/g) | -0.069 (0.074) | -0.029 (0.079) | -0.217 (0.076) | 0.034 (0.073)
Statistical Analysis 1: Comparison: BI 685509 1 mg TID vs BI 685509 2mg TID vs BI 685509 3 mg TID vs Placebo; A flat vs. non-flat dose-response relationship across the 3 doses of BI 685509 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (linear, exponential, quadratic, Emax and Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 0.050). The total daily dose was considered for MCP-Mod analysis (placebo, active BI 685509 3 mg, 6 mg, and 9 mg); Test type: Other — MMRM estimates were used as input for the MCP-Mod. including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit as well as random effects of patient; p = 0.0245, MCP-Mod exponential model fit; Model assumption: 20% of the maximum effect is achieved at 3 mg
Statistical Analysis 2: Comparison: BI 685509 1 mg TID vs BI 685509 2mg TID vs BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0294, MCP-Mod linear model fit; Model assumption: No assumption was needed
Statistical Analysis 3: Comparison: BI 685509 1 mg TID vs BI 685509 2mg TID vs BI 685509 3 mg TID vs Placebo; Test type: Other — A flat vs. non-flat dose-response relationship across the 3 doses of BI 685509 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (linear, exponential, quadratic, Emax and Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 0.050). The total daily dose was considered for MCP-Mod analysis (placebo, active BI 685509 3 mg, 6 mg, and 9 mg); p = 0.0468, MCP-Mod quadratic model fit — MMRM estimates were used as input for the MCP-Mod. including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit as well as random effects of patient; Model assumption: 50 % of the maximum effect is achieved at a dose of 3 mg. 90 % of the maximum effect is achieved at a dose of 6 mg
Statistical Analysis 4: Comparison: BI 685509 1 mg TID vs BI 685509 2mg TID vs BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0586, MCP-Mod Emax model fit; Model assumption: 80% of the maximum effect is achieved at 6 mg
Statistical Analysis 5: Comparison: BI 685509 1 mg TID vs BI 685509 2mg TID vs BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0659, MCP-Mod Sigmoid emax model fit; Model assumption: 30 % of the maximum effect is achieved at a dose of 3 mg. 90 % of the maximum effect is achieved at a dose of 6 mg
Statistical Analysis 6: Comparison: BI 685509 1 mg TID vs Placebo; Least Square Means difference and 95% confidence interval were estimated by restricted maximum likelihood based Mixed-effect Model for Repeated Measures ((REML)-based MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12 and Week 20) as well as random effects of patient; Test type: Other; p = 0.3224, Mixed-effect Model Repeat Measurement; Mean Difference (Net) = -0.103, 95% CI 2-sided [-0.309 to 0.102] — Least Squares Mean of "1 mg BI 685509 TID"- Least Squares Mean of"Placebo"
Statistical Analysis 7: Comparison: BI 685509 2mg TID vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = 0.5616, Mixed-effect Model Repeat Measurement; Mean Difference (Net) = -0.063, 95% CI 2-sided [-0.275 to 0.150] — Least Squares Mean of "2 mg BI 685509 TID"- Least Squares Mean of "Placebo"
Statistical Analysis 8: Comparison: BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = 0.0183, Mixed-effect Model Repeat Measurement; Mean Difference (Net) = -0.251, 95% CI 2-sided [-0.459 to -0.043] — Least Squares Mean of "3 mg BI 685509 TID"- Least Squares Mean of "Placebo"

2. Secondary Outcome: Change From Baseline in Log Transformed Urine Albumin Creatinine Ratio (UACR) Measured in First Morning Void Urine After 20 Weeks of Trial Treatment
Description: Change from baseline in log transformed Urine Albumin Creatinine Ratio (UACR) measured in First Morning Void urine after 20 weeks of trial treatment is reported. The first morning void (FMV) was the first urination after the patient woke up at their usual time to start their day. Least Square Means and Standard error were estimated by restricted maximum likelihood based Mixed-effect Model for Repeated Measures ((REML)-based MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12 and Week 20) as well as random effects of patient. The Least Squares Mean (Standard error) at Week 20 is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram/gram (mg/g)
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo
Number analyzed (Participants) | 57 | 53 | 56 | 56
milligram/gram (mg/g) | -0.112 (0.072) | -0.020 (0.076) | -0.258 (0.074) | 0.099 (0.072)
Statistical Analysis 1: Comparison: BI 685509 1 mg TID vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = 0.0396, Mixed Models Analysis; Mean Difference (Net) = -0.211, 0.95% CI 2-sided [-0.413 to -0.010] — Least Squares Mean of "1 mg BI 685509 TID"- Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: BI 685509 2mg TID vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = 0.2568, Mixed Models Analysis; Mean Difference (Net) = -0.120, 0.95% CI 2-sided [-0.327 to 0.088] — Least Squares Mean of "2 mg BI 685509 TID"- Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Net) = -0.357, 0.95% CI 2-sided [-0.560 to -0.154] — Least Squares Mean of "3 mg BI 685509 TID"- Least Squares Mean of "Placebo"

3. Secondary Outcome: Number of Patients Achieving UACR Decreases in 10-hour Urine of at Least 20% From Baseline After 20 Weeks of Trial Treatment
Description: Number of patients achieving Urine Albumin Creatinine Ratio (UACR) decreases in 10-hour urine of at least 20% from baseline after 20 weeks of trial treatment is reported. As soon as the First Morning Void sample was collected the clock starts for the 10-hour urine collection. During the 10-hour period every time the patient urinates, they collected their urine into a provided container. An aliquot of this urine was taken and used as the 10-hour UACR sample.
Time Frame: Baseline (day -14 and -7) and week 20 (day 141).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo
Number analyzed (Participants) | 57 | 53 | 56 | 56
Participants | 23 | 16 | 26 | 13
Statistical Analysis 1: Comparison: BI 685509 1 mg TID vs Placebo; Treatment, sodium-Glucose co-Transporter-2 Inhibitor (SGLT2i) use at baseline, and type of diabetes were used as covariates in the logistic regression model; Test type: Other; p = 0.0519, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.99 to 5.10] — Odds Ratio was calculated as BI 685509/ Placebo
Statistical Analysis 2: Comparison: BI 685509 2mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.4159, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.61 to 3.36] — Odds Ratio was calculated as BI 685509/ Placebo
Statistical Analysis 3: Comparison: BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0106, Regression, Logistic; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.28 to 6.55] — Odds Ratio was calculated as BI 685509/ Placebo

4. Secondary Outcome: Number of Patients Achieving UACR Decreases in First Morning Void Urine of at Least 20% From Baseline After 20 Weeks of Trial Treatment
Description: Number of patients achieving Albumin Creatinine Ratio (UACR) decreases in First Morning Void urine of at least 20% from baseline after 20 weeks of trial treatment. is reported. The first morning void (FMV) was the first urination after the patient woke up at their usual time to start their day.
Time Frame: Baseline (day -14 and -7) and week 20 (day 141).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3 mg TID | Placebo
Number analyzed (Participants) | 57 | 53 | 56 | 56
Participants | 23 | 13 | 29 | 11
Statistical Analysis 1: Comparison: BI 685509 1 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0176, Regression, Logistic; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.20 to 6.53] — Odds Ratio was calculated as BI 685509/ Placebo
Statistical Analysis 2: Comparison: BI 685509 2mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.5467, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.53 to 3.29] — Odds Ratio was calculated as BI 685509/ Placebo
Statistical Analysis 3: Comparison: BI 685509 3 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.91 to 10.39] — Odds Ratio was calculated as BI 685509/ Placebo

ADVERSE EVENTS:
Time Frame: From first BI 685509 intake until last BI 685509 intake or patient's trial termination date, whichever occurs earlier + 7 days of Residual effect period (REP), up to 148 days.
Description: Treated Set (TS): This set included all patients who were dispensed trial medication (BI 685509) and were documented to have taken at least 1 dose of open-label trial medication (BI 685509).
Groups:
- BI 685509 3mg TID: The patients were administered 1 milligram (mg) BI 685509 Film-coated tablets 3 times a day during the first 2 weeks of treatment, If the medication was tolerated, up-titration to 2 mg TID BI 685509 occurred after 2 weeks until Week 4 of treatment. Then if medication was tolerated, up-titration to 3 mg TID BI 685509 occurred from Week 5 until Week 20.
  The tablets were taken with water, with or without food. Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
Arm/Group | BI 685509 1 mg TID | BI 685509 2mg TID | BI 685509 3mg TID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 1/61 | 2/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 4/61 | 8/61 | 7/61 | 4/58
Other Adverse Events (participants affected / at risk) | 13/61 | 15/61 | 15/61 | 14/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 685509 1 mg TID (N=61) | BI 685509 2mg TID (N=61) | BI 685509 3mg TID (N=61) | Placebo (N=58)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1 | 0 | 0
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 685509 1 mg TID (N=61) | BI 685509 2mg TID (N=61) | BI 685509 3mg TID (N=61) | Placebo (N=58)
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 4
Oedema peripheral (General disorders) | 2 | 5 | 5 | 1
COVID-19 (Infections and infestations) | 2 | 3 | 3 | 3
Hypertension (Vascular disorders) | 3 | 2 | 3 | 6
Hypotension (Vascular disorders) | 3 | 6 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04750577/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04750577/SAP_001.pdf